CLINICAL TRIAL: NCT00712049
Title: Effects of Nicotinic Acid Plus Simvastatin Versus Simvastatin Alone on Carotid and Femoral Intima-Media Thickness in Patients With Peripheral Artery Disease (NASCIT)-A Randomized Controlled Trial
Brief Title: Effects of Nicotinic Acid Plus Simvastatin Versus Simvastatin Alone on Carotid and Femoral Intima-Media Thickness in Patients With Peripheral Artery Disease (NASCIT)
Acronym: NASCIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. Dr. Renate Koppensteiner, Medical University Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.0-2007
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Dyslipidemia; Atherosclerosis
Keywords: intima-media-thickness; dyslipidemia; progression of atherosclerosis; peripheral artery disease; major cardiovascular events
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis; Peripheral Arterial Disease | interventions — Simvastatin; Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Nicotinic acid + Simvastatin
  Interventions: Drug: simvastatin; Drug: Nicotinic Acid
- 2 (Active Comparator): Simvastatin
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: simvastatin — simvastatin 40 mg
Drug: Nicotinic Acid — daily dose starting with 500 mg, up to 2000mg
  Arms: 1

SUMMARY:
Dyslipidaemia is characterized by low plasma levels of high-density lipoprotein cholesterol (HDL-c), elevated triglycerides and an increase in low density lipoprotein (LDL-c) particles, and has been unequivocally established as a most important cardiovascular risk factor. While statins are effective in reducing plasma levels of LDL-c, these drugs have only modest effects on raising HDL-c (typically by less than 10%), even with aggressive statin therapy. However, increasing evidence suggests that low HDL-c might be at least as relevant as high LDL-c in promoting the development and progression of atherosclerosis. The beneficial effect of raising HDL-c on clinical outcome has already been demonstrated by several studies.

Nicotinic acid is the most potent agent available for raising plasma levels of HDL-c by up to 29% at clinically recommended doses, and substantially lowers triglycerides and LDL-c. Furthermore, nicotinic acid is also the most potent lipid lowering agent available that reduces Lp(a), an independent marker of cardiovascular risk. In a recent study patients with coronary artery disease had a 21% increase in HDL-c and a 13% decrease in triglycerides, and these beneficial effects on lipid status may have contributed to a stabilization or regression of carotid intima-media-thickness (IMT).The impact in patients with advanced atherosclerosis like peripheral artery disease (PAD) in unknown.

The investigators hypothesized that nicotinic acid in addition to statin therapy may inhibit progression of peripheral arterial atherosclerosis. Therefore, the aim of the present randomized controlled trial is to investigate the effects of nicotinic acid (daily dose starting with 500 mg, up to 2000mg) in addition to simvastatin (40 mg daily) versus simvastatin (40mg daily) monotherapy in patients with low serum HDL-C levels and PAD with respect to changes of carotid and femoral IMT, changes of patients´ lipid status and occurrence of major adverse cardiovascular events (MACE).

ELIGIBILITY:
Inclusion Criteria:

* PAD defined as an ABI ≤0.9 or >1.3 in patients with low serum HDL cholesterol levels (<45mg/dL in men, <55 mg/dL in women)

Exclusion Criteria:

* Elevated liver enzymes (above 2 times the normal level)
* Skeletal muscle myopathy or elevated serum CK levels
* Allergy or hypersensibility to either statins or nicotinic acid
* Women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-06

PRIMARY OUTCOMES:
change of carotid and femoral IMT from baseline to 6 and 12 months follow up and occurrence of major adverse cardiovascular events (MACE) | 6 and 12 months

SECONDARY OUTCOMES:
changes of grey scale median (GSM) score from baseline to follow-up, and changes of serum levels of total cholesterol, low-density lipoprotein cholesterol (LDL-c), high-density lipoprotein cholesterol (HDL-c), triglycerides and lipoprotein (a). | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Renate Koppensteiner, Prof. Dr., Principal Investigator — Division of Angiology, Department of Internal Medicine II, Medical University Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria